CLINICAL TRIAL: NCT04646317
Title: To Observe the Hemodynamic Stability of Dexmedetomidine in Hypertensive Patients Undergoing Laparoscopic Cholecystectomy.
Brief Title: Hemodynamic Stability of Dexmedetomidine in Hypertensive Patients Undergoing Laparoscopic Cholecystectomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Ruth K.M. Pfau Civil Hospital, Karachi (Other Government)
Responsible Party: Principal Investigator, Muhammad Imran Riasat, Senior Registerar, Dr. Ruth K.M. Pfau Civil Hospital, Karachi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PfauCHKarachi
Record Dates: First submitted 2020-10-24; First posted 2020-11-27 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Hypertension; Laparoscopic Cholecystectomy
Keywords: Attenuation; dexmedetomidine; pneumoperitoneum; hemodynamic stability; pressor response; laryngoscopy response; intubation response
MeSH Terms: conditions — Hypertension; Pneumoperitoneum | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Who Masked: Participant, Care Provider
Masking Description: Patients and care provider do not know about the interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine infusion four 50 ml syringes containing 1 microgram per ml dexmedetomidine
  Interventions: Drug: Dexmedetomidine injection
- normaL SALINE 0.9% (Placebo Comparator): Four 50 ml syringes of .9 % Normal SALINE
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine injection — Infusion of dexmedetomidine will be prepared in Four syringes of 50ml containing dexmedetomidine in concentration of 1 microgram per millilitre.
  Other Names: dexmedetomidine
  Arms: Dexmedetomidine
Drug: Normal Saline — 0.9% as placebo
  Arms: normaL SALINE 0.9%

SUMMARY:
Dexmedetomidine provides better hemodynamic stability to the patients with hypertension undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic surgeries form an essence of today's surgical practice because of its magnification, less cosmetic scar, less postoperative pain, and decreased hospital stay along with less morbidity and mortality.

According to the American Heart Association (AHA), approximately 86 million adults (34%) in the United States are affected by hypertension, which is defined as a systolic blood pressure (SBP) of 140 mm Hg or more or a diastolic blood pressure (DBP) of 90 mm Hg or more, taking anti-hypertensive medication of those with high blood pressure (BP), 78% were aware they were hypertensive, 68% were being treated with anti-hypertensive agents, and only 64% of treated individuals had controlled hypertension.

Anaesthetic management in these patients has become complicated due to cardiopulmonary changes occurring during creation of pneumoperitoneum with CO2 and patient position required for different laparoscopy surgeries. Effects of pneumoperitoneum for laparoscopic surgeries on heart rate and blood pressure was recognized more than 50years ago and the magnitude of the changes was observed to depend on the depth of anesthesia. The cardiovascular, neuroendocrine, and renal changes induced by the CO2 pneumoperitoneum produce a complex pathophysiological state remarkably similar to that in patients with chronic heart failure, though the initiating event is clearly very different. In normotensive subjects these hemodynamic changes are short lived5and probably of little significance. However, these haemodynamic alterations are hazardous to the patients with hypertension, myocardial insufficiency or cerebrovascular disease.

Various pharmacologic and nonpharmacological methods have been tried to limit the pressor response following the creation of pneumoperitoneum. The success rate is variable with different methods because each method has its own merits and demerits. In several clinical trials drugs like opioids, β-blockers, lidocaine, nitrate calcium channel blockers or magnesium have already been used orally or parenterally to obtund this sympathoadrenal response. Recently, there is considerable interest in the use of α2-adrenergic agonists to provide hemodynamic stability during pneumoperitoneum.

Dexmedetomidine famous for its awake sedation is eight times more selective than clonidine for the α2-adrenergic receptors. The ratio of α2:α1 activity of dexmedetomidine is 1620:1. It activates pro-survival kinases and attenuates ischemia and hypoxic injury, including cardio protection. Concurrent infusion during surgery reduces anesthetic consumption by 20-50% , and produces a decrease in heart rate and blood pressure that may be advantageous for hypertensives. Hypertension associated to pneumoperitoneum in normotensive patients has been controlled with the loading dose of dexmedetomidine. So our rational is to see the hemodynamic stability of dexmedatomindine in hypertensive patients undergoing pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients of both genders of age 17 years to 70 years who are undergoing laparoscopic cholecystectomy.
* ASA II and III

Exclusion Criteria:

* Patients with a prior history of cardiac disease like ischemic heart disease, valvular disorders, undergone previous valve replacements, infective endocarditis and rheumatic fever.
* Renal diseases like acute kidney injury and chronic renal diseases.
* Endocrinal diseases like pheochromocytoma, hyperthyroidism, hypothyroidism, cushing disease etc.
* Pregnant and lactating females
* Short thick neck with anticipated difficult intubation
* Any sort of obstructive restrictive or reactive airway disease
* Patient allergic to any of the study medications.
* Obese patients (BMI>35)
* Narcotic addicts

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2021-03-02 (Estimated); Study Completion 2021-03-02 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic blood pressure during pneumoperitoneum | From baseline to the end of pneumoperitonium, an average of 2 hours
  Systolic blood pressure will be noted on baseline, after induction, every 5 minutes after induction to the end of pneumoperitonium and every 5 minutes for 30 minutes post operatively
change in Diastolic blood pressure during pneumoperitoneum | from baseline to the end of pneumoperitoneum, an average of 2 hours
  Diastolic blood pressure will be noted on baseline, after induction, every 5 minutes after induction to the end of pneumoperitonium and every 5 minutes for 30 minutes post operatively
change in Mean Arterial blood pressure during pneumoperitoneum | from baseline to the end of pneumoperitoneum, an average of 2 hours
  Mean Arterial blood pressure will be noted on baseline, after induction, every 5 minutes after induction to the end of pneumoperitonium and every 5 minutes for 30 minutes post operatively
change in Heart Rate during pneumoperitoneum | from baseline to the end of pneumoperitoneum, an average of 2 hours
  Heart rate will be noted on baseline, after induction, every 5 minutes after induction to the end of pneumoperitonium and every 5 minutes for 30 minutes post operatively

SECONDARY OUTCOMES:
Systolic blood pressure intubation | Induction
  SBP will be noted at the induction.
Diastolic Blood pressure intubation | Induction
  DBP will be noted at the induction
Mean Arterial blood pressure intubation | Induction
  MAP will be noted at the induction.
heart rate intubation | Induction
  HR will be noted at the induction.
Post operative sedation | every 5 minutes, up to 30minutes
  Modified Ramsey score use for sedation, it consist of 1-6 where 6 indicates worst(no response) and 6 indicates good response From completion of surgery to 30 minutes post operatively
Post operative analgesia | every 5 minutes, up to 30minutes
  Visual analogue scale From completion of surgery to 30 minutes post operatively (0 no pain, 10 wost pain)
Complication | every 5 minutes from induction, up to 30 minutes post procedure
  bradycardia, tachycardia, hypertension and hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Imran, FCPS, Principal Investigator — Dow University of Health Sciences; Hanya Javaid, FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dr. Ruth K.M Pfau Civil Hospital Dow university of health sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No